CLINICAL TRIAL: NCT06753474
Title: Influenza Human Challenge Model Using H3N2 (A/Texas/71/2017 (H3N2), Clade 3C3a)
Brief Title: A/Texas Flu Challenge
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: NATIONAL PHILANTHROPIC TRUST (Unknown)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor of Medicine, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00008371
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Live Influenza Virus RG-A/Texas/71/2017 (H3N2 (Experimental): Participants will be pre-screened up to sixty days before the challenge study to identify baseline HAI titer. Participants will either be in the intranasal challenge or the natural exposure cohort.
  Interventions: Biological: Influenza Virus influenza A H3N2 strain

INTERVENTIONS:
Biological: Influenza Virus influenza A H3N2 strain — Live Influenza Virus RG-A/Texas/71/2017 (H3N2). It is a cell-grown, reverse genetics-derived influenza A virus manufactured to conduct clinical trials that involve controlled human infection with influenza A virus. This influenza human challenge virus was produced for the National Institute of Allergy and Infectious Diseases (NIAID).
  The final Drug Product Live Influenza Virus RG-A/Texas/71/2017 (H3N2) (Lot #1507-232149) vial contains 1.86 X 106 median tissue culture infectious doses (TCID50)/mL formulated in 1X sucrose-phosphate-glutamate (SPG; 7.4% sucrose, 3.8 mM KH2PO4, 7.2 mM K2HPO4, 5.4 mM L-glutamic acid) in Ex-Cellä 293 serum-free medium (Sigma-Aldrich). It is susceptible to the FDA-approved neuraminidase (NA) inhibitors (NAI) oseltamivir phosphate, zanamivir, and peramivir, and the polymerase acidic (PA) inhibitor (PAI) baloxavir marboxil.x
  Other Names: RG-A/Texas/71/2017 H3N2

SUMMARY:
This study is designed to help us better understand how the immune system responds to the flu and how flu is transmitted in the environment. The ultimate goal is to develop better vaccines and drugs to protect against or fight the flu.

This study will describe how the body's immune system responds to the flu virus during and after infection and how the flu virus is transmitted in the environment. The study will use a flu virus called A/Texas/71/2017 (H3N2), clade 3C3a produced specifically for clinical research in controlled conditions. The study will also assess the safety of the H3N2 influenza challenge in healthy participants. Mild to moderate symptoms are expected based on previous studies with this strain of influenza.

Study volunteers will be recruited and screened from the general population of metro Atlanta through advertisements or identified from a database of research participants who have previously agreed to be contacted for future research studies. Participants will provide written consent before study participation.

Up to 200 healthy adults, 18-49 years old, will be screened for participation. Eligible participants will take part in the study over 5 months. Enrolled participants will be admitted to Emory University Hospital during which time they will receive the influenza virus in the form of a spray in the nose or exposure to infected participants followed by an 8-12 day inpatient stay for observation. Follow-up outpatient visits will take place at the Hope Clinic of the Emory Vaccine Center. Participants will receive compensation (pro-rated for all visits completed) for their time and effort. There will be no costs to participants as a result of being in the study.

DETAILED DESCRIPTION:
Influenza A continues to circulate widely in the human population and causes significant morbidity and mortality. Current vaccines have variable effectiveness year-to-year, with observable breakthrough infections each season, and have limited effectiveness in certain at-risk members of the population. Although basic and clinical influenza research has broadened our understanding of viral immunology, transmission, and pathogenesis, important questions, particularly concerning correlates of protection, viral evolution, and transmission, remain unanswered. Many of these questions can only be approached through studies in humans.

As more broadly protective vaccines are developed, efficient and comprehensive methods of determining their value will be imperative. One of the key components and gap-filling measures in the National Institute of Allergy and Infectious Diseases (NIAID) strategic plan for universal influenza vaccines is to expand our capacity to conduct human challenge studies with relevant influenza challenge viruses to facilitate early evaluation of new vaccines and to further our understanding of flu pathogenesis and immunity. The goal of this study is to conduct a human challenge study to build upon our success at establishing the influenza challenge model at Emory to better understand influenza pathogenesis, immunity, transmission, and evolution using an H3N2 challenge stock.

Human challenge studies for influenza are a particularly attractive modality for the development of a universal influenza vaccine. As outlined by NIAID's strategic plan, a universal flu vaccine would be at least 75% effective, maintain protection for at least one year, protect against group I (e.g., H1, H5) and II (e.g., H3, H7) influenza A virus strains, and be effective for all age groups. ix The strategic plan also states that a human challenge model could offer unique benefits to better understand the concept of imprinting, determine correlates of protection against influenza, and evaluate different universal influenza vaccine candidates. The development of universal vaccine strategies that reduce transmission potential and can protect from infection by aerosolized viruses will be a strategic advantage for reducing the public health burden from influenza viruses.

ELIGIBILITY:
Inclusion Criteria:

* Can understand and comply with all planned study procedures.
* Healthy, non-pregnant, non-breast-feeding persons aged ≥18 and ≤49 years of age inclusive at the time of challenge.
* Persons biologically able to become pregnant must be practicing abstinence or using an acceptable method of birth control for at least 30 days before the challenge through the duration of the trial. Persons biologically able to make someone pregnant must agree not to get their partner pregnant for the duration of the trial.

  * A person is considered of childbearing potential unless post-menopausal (absence of menses for ≥1 year) or surgically sterilized (tubal ligation/salpingectomy, bilateral oophorectomy, or hysterectomy).
  * Acceptable contraception methods for persons of childbearing potential include but are not limited to: sexual abstinence from intercourse with partners biologically able to make them pregnant, monogamous relationship with a vasectomized partner, barrier methods such as condoms or diaphragms with spermicide or foam, effective devices (IUDs, NuvaRing®) or licensed hormonal products such as implants, injectables or oral contraceptives.
* Persons of childbearing potential must have a negative serum or urine pregnancy test at screening and a negative urine pregnancy test within 24 hours before challenge.
* Are in good general health, as determined by the study investigator within 30 days of challenge, and do not have any of the following conditions:

  * Chronic pulmonary disease (e.g., asthma or emphysema).
  * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
  * Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
  * Immunosuppression, ongoing malignancy, or history of malignancy (excluding non-melanotic skin cancer in remission without treatment for more than 5 years).
  * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
  * History of postinfectious or postvaccine neurological sequelae.
  * Autoimmune, inflammatory, vasculitis, or rheumatic disease, including but not limited to systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma.
* Demonstrate knowledge and comprehension of the study by scoring ≥70% on a quiz on the study protocol and policies.
* Agrees to not use cigarettes, e-cigarettes, marijuana, or other tobacco products during the quarantine period.
* Agrees not to use prescription or over-the-counter medications that could impact influenza challenge efficacy or symptoms (including oseltamivir, zanamivir, peramivir, baloxavir marboxil, amantadine and rimantadine, aspirin, intranasal steroids, acetaminophen, decongestants, antihistamines, and other NSAIDs), within 14 days before challenge and through the quarantine period, unless approved by the investigator.

Exclusion Criteria:

* Have household contact with or have daily contact with:

  * Children under 5 years of age.
  * Children and/or teenagers who are receiving long-term aspirin therapy.
  * Persons who are pregnant or who are trying to become pregnant.
  * Persons older than 65 years of age.
  * Persons of any age with significant chronic medical conditions such as:

    * Chronic pulmonary disease (e.g., asthma, emphysema, COPD).
    * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
    * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic metabolic disease (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
    * Immunosuppression or cancer.
    * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
* Healthcare workers with patient contact during the two weeks following the influenza challenge.
* Plan to live in a confined environment (e.g., ship, camp, or dormitory) during the two weeks following the influenza challenge.
* Pregnant persons or are planning to become pregnant at any time during the study.
* Persons who are breastfeeding or plan to breastfeed at any time during the study.
* Have a body mass index (BMI) less than or equal to 18.5 or greater than or equal to 35.
* Smoke more than four cigarettes, e-cigarettes, marijuana, or other tobacco products weekly within 60 days before the challenge.
* Have moderate or severe illness within seven days before the challenge. This includes but is not limited to an oral temperature of ≥100°F, diarrhea, or vomiting.
* Have a pulse rate of less than 55 beats per minute (bpm) or greater than 100 bpm (participants will not be excluded if the heart rate is 55 bpm with moderate exercise (e.g., walking up two flights of stairs))
* Have a systolic blood pressure of less than 90 mmHg or greater than 140 mmHg on two separate measurements (screening and pre-challenge).
* Have a diastolic blood pressure of less than 50 mmHg or greater than 90 mmHg on two separate measurements (screening and pre-challenge).
* Have long-term (≥2 weeks) use of high-dose oral (≥20 mg per day prednisone or equivalent) or parenteral glucocorticoids, or high-dose inhaled steroids for greater than 7 days in the last 3 months.
* Have an active HIV, hepatitis B, or hepatitis C infection.
* Have screening laboratory test results (white blood cells [WBC], absolute neutrophil count [ANC], hemoglobin, platelets) that are outside the laboratory reported normal values and deemed clinically significant by the study investigator.
* Have a serum creatinine greater than 1.1 x upper limit of normal (ULN).
* Have an alanine aminotransferase (ALT) greater than 1.1 x ULN.
* Have abnormal findings on screening electrocardiogram deemed clinically significant by the study investigator.
* Have abnormal findings on screening chest X-ray deemed clinically significant by the study investigator.
* Have ongoing drug or alcohol abuse and/or dependence within five years of challenge.
* Have positive urine/serum test for drugs of abuse (i.e. cocaine, benzodiazepines, opiates, or metabolites).

Positive results for tetrahydrocannabinol (THC) will not be considered exclusionary. Metabolites and amphetamines as prescribed for a documented medical condition will also not be considered exclusionary.

* Have any medical, psychiatric, occupational, or behavioral problems that could make it difficult for the participant to comply with the protocol as determined by the investigator.
* Have received experimental products within 30 days before the challenge or plan to receive experimental products at any time during the study.
* Plan to enroll in another clinical trial that could interfere with the safety assessment of the investigational product at any time during the study period, including study interventions such as drugs, biologics, or devices.
* Plan to donate blood during the study.
* Have received a live vaccine within 30 days before the challenge or plan to receive a live vaccine before Day 31 post-challenge.
* Have received an inactivated vaccine within 14 days before the challenge or plan to receive an inactivated vaccine before Day 14 of the challenge.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mild to moderate influenza disease | Up to Day 12
  Number of participants with mild to moderate influenza disease (MMID) from challenge through discharge from quarantine.
Number of Serious Adverse Events | Up to Week 12
  The number of serious adverse events during the duration of the study will be evaluated.
Number of Participants with Severe Influenza Disease | Up to Day 12
  The number of participants experiencing severe influenza disease (MMID) from challenge to discharge from quarantine

SECONDARY OUTCOMES:
Change in Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HAI) | Baseline, Day 28
  The GMT of HAI to the challenge H3N2 strain will be evaluated.
Change in Geometric Mean Fold Rise (GMFR) of HAI | Baseline, Day 28
  The GMFR of HAI to the challenge H3N2 strain will be evaluated.
Change in Number of Participants with 4-fold Rise in HAI | Baseline, Day 28
  The number of participants with a 4-fold rise in HAI will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia
  - Hope Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available for sharing including data on safety, participant demographics, and immunogenicity.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available for sharing one year after the results from this study are published.
Access Criteria: Data will be made available for sharing with researchers who provide a methodologically sound protocol, to achieve the aims stated in the protocol. The proposal should be directed to nroupha@emory.edu. Requestors will need to sign a data access agreement.